CLINICAL TRIAL: NCT07096856
Title: Post Market Clinical Study to Evaluate the Performance of the Versius Surgical System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CMR Surgical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-00583
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cholecystectomy, Robotic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Robotic-Assisted Cholecystectomy Using the Versius Surgical System (Experimental)
  Interventions: Device: Robotic assisted cholecystectomy

INTERVENTIONS:
Device: Robotic assisted cholecystectomy — Robotic assisted cholecystectomy

SUMMARY:
The goal of this clinical trial is to learn how the Versius Surgical System, a robotic surgery device, works for gallbladder removal surgery (cholecystectomy) in adults. The main questions it aims to answer are:

How often can the surgery be successfully completed using Versius without needing to switch to a different surgical method?

What serious complications, if any, occur within 30 days after surgery?

Researchers will collect information from adult patients who have gallbladder surgery using the Versius system in U.S. hospitals. The purpose is to better understand how the device performs and how patients recover after surgery.

Participants will:

Be adults age 22 or older who are eligible for minimally invasive gallbladder surgery

Undergo robotic-assisted surgery using the Versius Surgical System

Allow the research team to collect data during surgery and up to 30 days after

Complete standard follow-up visits after discharge

Patients with certain medical conditions, such as cancer, high BMI (≥40 kg/m²), or contraindications to anesthesia or robotic surgery, will not be included in the study.

This study is sponsored by CMR Surgical Ltd., the manufacturer of the Versius system.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients 22 years of age and older, eligible for soft tissue minimal access surgery, for cholecystectomy 2. Patients providing written informed consent to participate in the study

Exclusion Criteria:

1. Patient unwilling to provide informed consent
2. Patients undergoing surgery or treatment for malignant disease
3. Patients undergoing a concomitant surgical procedure
4. Medical contraindication for general anaesthesia or minimally invasive procedure
5. Contraindication for undergoing surgery with Versius (Bleeding diathesis, Active pregnancy or BMI ≥40 kg/m2)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of successful completion of the cholecystectomy surgical procedure without unplanned conversions to open or other minimally invasive surgery | From start of surgery to end of procedure
  Rate of successful completion of the cholecystectomy surgical procedure without unplanned conversions to open or other minimally invasive surgery
Rate of serious adverse events up to 30 days post procedure. | From end of surgery through 30 days post-procedure
  Rate of serious adverse events up to 30 days post procedure.